CLINICAL TRIAL: NCT00201890
Title: DELTA - A Randomized Trial of Decongestive Lymphatic Therapy for Lymphedema in Women With Breast Cancer
Brief Title: Trial of Decongestive Lymphatic Therapy for Lymphedema in Women With Breast Cancer "DELTA STUDY"
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ontario Clinical Oncology Group (OCOG) (Other)
Collaborators: Canadian Breast Cancer Research Alliance (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CBCRA- 013260
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2012-10-10 (Estimated); Status verified 2012-10

CONDITIONS: Breast Cancer; Lymphedema
Keywords: Breast Cancer; Lymphedema; Treatment; Massage; Randomized; DLT therapy; Quality of Life; Decongestive Therapy; Breast Cancer related Lymphedema
MeSH Terms: conditions — Breast Neoplasms; Lymphedema; Breast Cancer Lymphedema | interventions — Gloves, Protective

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Standard of Care plus Lymphatic massage (Decongestive Lymphatic Therapy)
  Interventions: Procedure: Lymphatic Massage (Decongestive Lymphatic Therapy) (Arm 1)
- 2 (No Intervention): Standard of Care

INTERVENTIONS:
Procedure: Lymphatic Massage (Decongestive Lymphatic Therapy) (Arm 1) — 20 weeks of lymphatic massage therapy by a certified LMT in the Vodder technique Elastic Compression Sleeve and GLove
  Other Names: Elastic Compression Sleeeve and Glove (Arm 2)
  Arms: 1

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety and impact on quality of life of decongestive lymphatic therapy (DLT) in women who have completed treatment for breast cancer and present with lymphedema.

This is a multicentre trial enrolling 100 patients randomized to receive conservative care for arm lymphedema (Canadian Guidelines) with or without decongestive lymphatic therapy performed by a professional who has received training and certification in the technique of lymphatic draining massage.

Duration: One year after the last patient is randomized.

DETAILED DESCRIPTION:
Randomized patients receive either standard of care or standard of care plus DLT (five massage sessions per week for 4 consecutive weeks). Primary evaluation of all patients is recorded six weeks after randomization by measuring the affected limb and comparing with the unaffected one. There is an extended follow-up of one year.

ELIGIBILITY:
Inclusion Criteria:

* Women with a histological diagnosis of breast cancer experiencing edema in the ipsilateral arm such that there is a minimum 15% increase in arm volume over the opposite arm.
* Patients must have completed all primary and adjuvant treatments (surgery, chemotherapy, radiotherapy) prior to randomization. This is to ensure that scheduling difficulties with daily treatments do not arise. Patients may be currently taking tamoxifen or similar hormonal treatment.

Exclusion Criteria:

* Clinical or radiological evidence of active disease, either local or metastatic.
* History of contralateral cancer, axillary surgery, radiation or bilateral arm edema. (Edema volume will be taken as the increase in volume compared to the unaffected arm; previous therapy in the opposite arm will reduce the accuracy of measuring excess volume related to lymphedema.)
* Previous surgery involving nodal dissection or radiotherapy to other major node-bearing areas in the body such as the mediastinum or pelvis. Disruption of lymphatic flow in these potentially alternate routes may be compromised by such interventions. Patients are eligible after a simple hysterectomy (+/- oophorectomy).
* Previously undergone massage therapy for arm edema, or has used compression sleeve within the last month.
* Serious non-malignant disease, such as renal or cardiac failure, which would preclude daily treatment and follow up.
* Patients for whom massage is contraindicated, such as those with untreated infections or thromboses in the affected arm.
* Unable to commence therapy within 7 days of randomization.
* Psychiatric or addictive disorders which preclude obtaining informed consent or adherence to the protocol.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2003-03; Primary Completion 2009-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Percent reduction in excess arm volume as calculated from circumferential arm measurements | at 6 weeks

SECONDARY OUTCOMES:
Measurement of arm function | Midtreatment,6,12 24,52 weeks
Quality of life | Midtreament, 6 12,24,52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ian Dayes, MD, Study Director — Ontario Clinical Oncology Group (OCOG); Tim Whelan, MD, Principal Investigator — McMaster University; Jim Julian, M. Math, Principal Investigator — McMaster University; Lyn Kligman, RN, Principal Investigator — London Regional Cancer Centre; Kathy Pritchard, MD, Principal Investigator — Sunnybrook Regional Cancer Centre
Locations (9):
- Canada (9):
  - Cross Cancer Institute, Edmonton, Alberta
  - Dr. Leon Richard Oncology Centre, Moncton, New Brunswick
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Dr. H. Bliss Murphy Cancer Centre, St. John's, Newfoundland and Labrador
  - Juravinski Cancer Centre, Hamilton, Ontario
  - London Regional Cancer Centre, London, Ontario
  - Thunder Bay Regional Health Science Centre, Regional Cancer Centre, Thunder Bay, Ontario
  - Sunnybrook Regional Cancer Centre, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario